CLINICAL TRIAL: NCT00511355
Title: A Randomized, Open-Label, Comparative, Multi -Center Trial to Evaluate the Effects on Hemostasis, Lipids and Carbohydrate Metabolism, and on Adrenal and Thyroid Function of a Monophasic COC Containing 2.5 mg NOMAC and 1.5 mg E2 Compared to a Monophasic COC Containing 150 ug LNG and 30 ug EE
Brief Title: Effects on Hemostasis, Lipids, Carbohydrate Metabolism, Adrenal & Thyroid Function of the Combined Oral Contraceptive NOMAC-E2 Compared to a COC Containing LNG-EE (292004)(COMPLETED)(P05764)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05764; Organon Protocol No. 292004
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Nomegestrol Acetate (NOMAC) and Estradiol (E2), 2.5 mg NOMAC and 1.5 mg E2 monophasic combined oral contraceptive
  Interventions: Drug: NOMAC-E2
- LNG-EE (Active Comparator): Levonorgestrel and Ethinyl Estradiol Tablets (LNG-EE), 150 mcg LNG and 30 mcg EE
  Interventions: Drug: Levonorgestrel and Ethinyl Estradiol

INTERVENTIONS:
Drug: NOMAC-E2 — Nomegestrol Acetate and Estradiol (NOMAC-E2) Tablets, 2.5 mg NOMAC and 1.5 mg E2 taken once daily from Day 1 of menstrual period up to and including Day 28 for 6 consecutive 28-day cycles.
  Other Names: SCH 900121; Org 10486-0 (NOMAC); Org 2317 (E2)
  Arms: NOMAC-E2
Drug: Levonorgestrel and Ethinyl Estradiol — Levonorgestrel and Ethinyl Estradiol (LNG-EE) Tablets, 150 mcg LNG and 30 mcg EE taken once daily from Day 1 of menstrual period up to and including Day 28 for 6 consecutive 28-day cycles.
  Arms: LNG-EE

SUMMARY:
The primary purpose of this study is to evaluate the effects of the combined oral contraceptive (COC) NOMAC-E2 on hemostasis, lipids, carbohydrate metabolism, adrenal function, and thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women, at risk for pregnancy and not planning to use during trial medication use;
* Women in need for contraception and willing to use an oral contraceptive (OC) for 6 months (6 cycles);
* At least 18 but not older than 50 years of age at the time of screening;
* Body mass index = 17 and = 29 kg/m^2;
* Good physical and mental health;
* Willing to give informed consent in writing

Exclusion Criteria:

* Present use or use within 2 months prior to screening of any other hormonal treatment including sex hormones (other than contraceptives), insulin, thyroid and corticosteroid hormones (with the exception for local dermatological use);
* Contraindications for contraceptive steroids
* Presence or history (within 1 year before screening) of alcohol or drug abuse as judged by the (sub)investigator.
* An abnormal cervical smear (i.e.: dysplasia, cervical intraepithelial neoplasia [CIN], SIL, carcinoma in situ, invasive carcinoma) at screening or documentation of an abnormal smear performed within 6 months before screening;
* Clinically relevant abnormal laboratory result at screening as judged by the (sub) investigator;
* Use of an injectable hormonal method of contraception prior to screening; within 6 months of an injection with a 3 -month duration, within 4 months to screening of an injection with a 2-month duration, within 2 months of an injection with a 1-month duration;
* Before spontaneous menstruation has occurred following a delivery or abortion;
* Breastfeeding or within 2 months after stopping breastfeeding prior to the start of trial medication;
* Present use or use within 2 months prior to the start of the trial medication of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, lipid-lowering drugs, anticoagulants and herbal remedies containing Hypericum perforatum (St John's Wort);
* Use of pharmacological agents which affect the hemostatic system during the pretreatment blood sampling: vitamin K (only prohibited within two weeks prior to sampling), nonsteroidal anti-inflammatory drugs (NSAIDS) and aspirin (both only prohibited during the week prior to sampling);
* Administration of investigational drugs and/or participation in another clinical trial within 2 months prior to the start of the trial medication or during the trial period.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Result] Agren UM, Anttila M, Maenpaa-Liukko K, Rantala ML, Rautiainen H, Sommer WF, Mommers E. Effects of a monophasic combined oral contraceptive containing nomegestrol acetate and 17beta-oestradiol compared with one containing levonorgestrel and ethinylestradiol on haemostasis, lipids and carbohydrate metabolism. Eur J Contracept Reprod Health Care. 2011 Dec;16(6):444-57. doi: 10.3109/13625187.2011.604450. PMID 22066891

RESULTS

PARTICIPANT FLOW:
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 6 consecutive 28-day cycles.
- LNG-EE: Monophasic combined oral contraceptive (COC) tablets containing 0.150 mg levonorgestrel (LNG) and 0.030 mg
  ethinylestradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28 placebo tablets) for 6 consecutive 28-day cycles.
Period: Overall Study
Arm/Group | NOMAC-E2 | LNG-EE
Started | 60 | 61
Completed | 53 | 52
Not Completed | 7 | 9
Not completed — Adverse Event | 4 | 4
Not completed — Pregnancy Wish | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other Reason | 0 | 1
Not completed — Pre-treatment (serious) adverse event | 0 | 1
Not completed — Withdrawal of informed consent | 0 | 1
Not completed — Other reason pre-treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- NOMAC-E2: All-participants-treated group. Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 6 consecutive 28-day cycles
- LNG-EE: All-participants-treated group. Monophasic combined oral contraceptive (COC) tablets containing 0.150 mg levonorgestrel (LNG) and 0.030 mg
  ethinylestradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 6 consecutive 28-day cycles
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | LNG-EE | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] — All-participants-treated group. For the LNG-EE arm, this population excludes 3 subjects who were randomized but not treated.
  years | 28.2 (8.2) | 29.1 (7.8) | 28.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants] — All-participants-treated group. For the LNG-EE arm, this population excludes 3 subjects who were randomized but not treated.
  Participants
    Female | 60 | 58 | 118
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Prothrombin Fragments 1 + 2
Description: Serum samples were obtained under fasting conditions (no food or alcoholic beverages within 12 hours of serum sampling). Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: All-participants-treated group; n = number of participants with non-missing baseline value and non-missing change from baseline to Cycle 6
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 0.18 (0.20) | 0.19 (0.08)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 0.31 (1.06) | 0.42 (1.17)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0849, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

2. Primary Outcome: Serum Concentration of D-Dimer
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L Fibrinogen Equivalent Units (FEU)
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mg/L Fibrinogen Equivalent Units (FEU)
  Baseline (n=60; NOMAC-E2; n=58) | 0.21 (0.16) | 0.19 (0.14)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 0.18 (0.14) | 0.26 (0.21)

3. Primary Outcome: Activated Protein C (APC) Resistance Ratio (Endogenous Thrombin Potential [ETP]-Based)
Description: Serum samples were obtained under fasting conditions (no food or alcoholic beverages within 12 hours of serum sampling). APC resistance ratio (ETP-based) measures the anticoagulation response of plasma to APC after activation of the extrinsic coagulation pathway. An increase in the ratio indicates a reduced responsiveness to APC. Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Ratio
  Baseline (n=59 NOMAC-E2; n=58 LNG-EE) | 0.80 (0.33) | 0.83 (0.40)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 1.14 (0.45) | 1.99 (0.76)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

4. Primary Outcome: Serum Concentration of Clotting Factor VIIa
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
U/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 84 (32) | 85 (37)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 118 (180) | 98 (66)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.4191, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

5. Primary Outcome: Serum Concentration of Clotting Factor VIIc
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 105 (24) | 105 (22)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 109 (31) | 96 (25)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

6. Secondary Outcome: Serum Concentration of Total Testosterone
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60, NOMAC-E2; n=58 LNG-EE) | 1.68 (0.75) | 1.90 (0.94)
  Cycle 6 (n=53, NOMAC-E2; n=52 LNG-EE) | 1.23 (0.86) | 0.91 (0.57)

7. Secondary Outcome: Serum Concentration of Free Testosterone
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
pmol/L
  Baseline (n=60, NOMAC-E2; n=58 LNG-EE) | 24.5 (14.9) | 26.3 (16.6)
  Cycle 6 (n=53, NOMAC-E2; n=52 LNG-EE) | 12.8 (8.8) | 9.9 (6.7)

8. Secondary Outcome: Serum Concentration of Dehydroepiandrosterone Sulphate (DHEAS)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
umol/L
  Baseline (n=60, NOMAC-E2; n=58 LNG-EE) | 4.94 (2.24) | 5.19 (2.26)
  Cycle 6 (n=53, NOMAC-E2; n=52 LNG-EE) | 4.32 (1.82) | 4.00 (1.91)

9. Primary Outcome: Serum Concentration of Clotting Factor VIII
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 93 (32) | 95 (32)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 89 (34) | 98 (30)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.3779, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

10. Primary Outcome: Serum Concentration of Clotting Factor II
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 94 (11) | 94 (12)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 95 (13) | 97 (11)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.5027, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

11. Primary Outcome: Serum Concentration of Antithrombin III
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 100 (10) | 99 (11)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 102 (9) | 96 (12)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0041, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

12. Primary Outcome: Serum Concentration of Protein S (Free)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 85 (16) | 86 (14)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 99 (20) | 99 (17)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.9662, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

13. Primary Outcome: Serum Concentration of Protein S (Total)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 78 (12) | 79 (10)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 83 (12) | 76 (9)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

14. Primary Outcome: Serum Concentration of Protein C
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of normal
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of normal
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 107 (18) | 103 (19)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 108 (21) | 113 (20)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

15. Primary Outcome: APC Resistance Ratio (Activated Partial Thromboplastin Time [APTT]-Based)
Description: Serum samples were obtained under fasting conditions (no food or alcoholic beverages within 12 hours of serum sampling). APC resistance ratio (APTT-based) measures the anticoagulation response of plasma to APC after activation of the intrinsic coagulation pathway. An increase in the ratio indicates a increased responsiveness to APC. Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Ratio
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 1.01 (0.13) | 1.00 (0.13)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 1.05 (0.13) | 1.03 (0.12)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.9662, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

16. Primary Outcome: Serum Concentration of Sex Hormone Binding Globulin (SHBG)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 74 (34) | 77 (26)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 108 (44) | 100 (31)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0187, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

17. Primary Outcome: Serum Concentration of C-Reactive Protein (CRP)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mg/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 0.82 (1.16) | 0.98 (1.35)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 1.32 (2.36) | 4.43 (8.43)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

18. Primary Outcome: Serum Concentration of Total Cholesterol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 4.48 (0.87) | 4.53 (0.82)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 4.51 (0.83) | 4.48 (0.75)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.6886, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

19. Primary Outcome: Serum Concentration of High Density Lipoprotein (HDL)-Cholesterol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 1.63 (0.36) | 1.68 (0.33)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 1.65 (0.34) | 1.41 (0.26)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

20. Primary Outcome: Serum Concentration of HDL2-cholesterol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=58 NOMAC-E2; n=50 LNG-EE) | 0.63 (0.26) | 0.69 (0.29)
  Cycle 6 (n=52 NOMAC-E2; n=51 LNG-EE) | 0.55 (0.25) | 0.40 (0.18)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

21. Primary Outcome: Serum Concentration of HDL3-cholesterol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=58 NOMAC-E2; n=50 LNG-EE) | 1.10 (0.16) | 1.14 (0.19)
  Cycle 6 (n=52 NOMAC-E2; n=51 LNG-EE) | 1.16 (0.16) | 1.10 (0.14)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0083, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

22. Primary Outcome: Serum Concentration of Low Density Lipoprotein (LDL)-Cholesterol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 2.41 (0.73) | 2.47 (0.66)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 2.40 (0.71) | 2.61 (0.74)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0455, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

23. Primary Outcome: Serum Concentration of Apolipoprotein A-1
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
g/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 1.58 (0.27) | 1.60 (0.25)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 1.78 (0.27) | 1.67 (0.20)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

24. Primary Outcome: Serum Concentration of Apolipoprotein B
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
g/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 0.64 (0.17) | 0.64 (0.15)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 0.68 (0.17) | 0.80 (0.21)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

25. Primary Outcome: Serum Concentration of Lipoprotein(a)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
g/L
  Baseline (n=60 NOMAC-E2; n=57 LNG-EE) | 0.15 (0.18) | 0.15 (0.14)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 0.17 (0.22) | 0.12 (0.11)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

26. Primary Outcome: Serum Concentration of Total Triglycerides
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 0.94 (0.30) | 0.82 (0.23)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 1.00 (0.37) | 1.02 (0.32)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0078, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

27. Primary Outcome: Area Under the Curve Over 3 Hours (AUC3) for Glucose (Oral Glucose Tolerance Test [OGTT])
Description: Blood glucose levels were determined as fasting values just before oral glucose intake and each half hour thereafter for 2 hours and again after 3 hours. Oral glucose tolerance was analysed using the (unadjusted) area under the curve over the 3 hours (AUC3). Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hrs*mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
hrs*mmol/L
  Baseline (n=59 NOMAC-E2; n=55 LNG-EE) | 15.82 (3.27) | 14.44 (2.47)
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 16.09 (3.05) | 16.69 (3.15)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

28. Primary Outcome: Incremental AUC3 for Glucose (OGTT)
Description: Blood glucose levels were determined as fasting values just before oral glucose intake and each half hour thereafter for 2 hours and again after 3 hours. Oral glucose tolerance was analysed using the (unadjusted) area under the curve over the 3 hours (AUC3). Incremental area under the curve was defined as incremental AUC3 = AUC3 - 3*fasting concentration. Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hrs*mmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
hrs*mmol/L
  Baseline (n=59 NOMAC-E2; n=55 LNG-EE) | 1.58 (3.05) | 1.06 (2.55)
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 1.76 (2.72) | 3.19 (3.03)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

29. Primary Outcome: AUC3 for Insulin (OGTT)
Description: Blood insulin levels were determined as fasting values just before oral glucose intake and each half hour thereafter for 2 hours and again after 3 hours. Oral glucose tolerance was analysed using the (unadjusted) area under the curve over the 3 hours (AUC3). Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hrs*pmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
hrs*pmol/L
  Baseline (n=51 NOMAC-E2; n=50 LNG-EE) | 650 (298) | 558 (182)
  Cycle 6 (n=46 NOMAC-E2; n=47 LNG-EE) | 658 (281) | 721 (264)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

30. Primary Outcome: Incremental AUC3 for Insulin (OGTT)
Description: Blood insulin levels were determined as fasting values just before oral glucose intake and each half hour thereafter for 2 hours and again after 3 hours. Oral glucose tolerance was analysed using the (unadjusted) area under the curve over the 3 hours (AUC3). Incremental area under the curve was defined as incremental AUC3 = AUC3 - 3*fasting concentration. Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hrs*pmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
hrs*pmol/L
  Baseline (n=51 NOMAC-E2; n=50 LNG-EE) | 517 (268) | 451 (160)
  Cycle 6 (n=46 NOMAC-E2; n=47 LNG-EE) | 534 (239) | 603 (237)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.0024, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

31. Primary Outcome: Serum Concentration of Hemoglobin Type A1c (HbA1c)
Description: Serum samples were obtained under fasting conditions (no food or alcoholic beverages within 12 hours of serum sampling). HbA1c was determined before glucose loading. Each cycle consists of 28 days.
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
Percent of glycosylated hemoglobin
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 5.3 (0.3) | 5.3 (0.2)
  Cycle 6 (n=53 NOMAC-E2; n=51 LNG-EE) | 5.3 (0.2) | 5.4 (0.2)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.3653, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

32. Primary Outcome: Serum Concentration of Total Cortisol
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 482 (128) | 502 (153)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 608 (167) | 944 (183)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

33. Primary Outcome: Serum Concentration of Corticosteroid Binding Globulin (CBG)
Description: as for outcome 1
Time Frame: Baseline to Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 910 (201) | 932 (163)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 1116 (252) | 1980 (389)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

34. Primary Outcome: Serum Concentration of Thyroid Stimulating Hormone (TSH)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mU/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 2.69 (1.28) | 2.20 (1.08)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 2.96 (2.05) | 2.75 (3.36)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.5668, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

35. Primary Outcome: Serum Concentration of Free Thyroxine (T4)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
pmol/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 14.0 (1.5) | 14.1 (1.5)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 15.9 (2.0) | 15.7 (2.1)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p = 0.1770, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

36. Primary Outcome: Serum Concentration of Thyroxin Binding Globulin (TBG)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
mg/L
  Baseline (n=60 NOMAC-E2; n=58 LNG-EE) | 20.3 (2.9) | 20.3 (3.3)
  Cycle 6 (n=53 NOMAC-E2; n=52 LNG-EE) | 24.2 (3.6) | 28.4 (5.3)
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; P-value compares the change from baseline to Cycle 6 between treatment groups; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — No correction for multiple testing was made; Cochran-Mantel-Haenszel test adjusted for age class applied on the changes from baseline

37. Secondary Outcome: Serum Concentration of Androstenedione
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60, NOMAC-E2; n=58 LNG-EE) | 9.60 (3.45) | 10.27 (3.91)
  Cycle 6 (n=53, NOMAC-E2; n=52 LNG-EE) | 8.23 (3.01) | 6.96 (3.37)

38. Secondary Outcome: Serum Concentration of Dihydrotestosterone (DHT)
Description: as for outcome 1
Time Frame: Baseline and Cycle 6 (between Days 15 and 21 of the cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 60 | 58
nmol/L
  Baseline (n=60, NOMAC-E2; n=58 LNG-EE) | 0.59 (0.21) | 0.62 (0.26)
  Cycle 6 (n=53, NOMAC-E2; n=52 LNG-EE) | 0.53 (0.28) | 0.36 (0.19)

39. Secondary Outcome: Number of In-treatment Pregnancies (With +2 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a maximum of 2 days. Each 13 cycles (28 days per cycle) constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 6 cycles
Population: The "restricted ITT" set included all participants treated and excluded nonpregnant participants who didn't have >=1 cycle expected to be at risk for pregnancy (with recorded use of condoms or w/o sexual intercourse per diary card data).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: Woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 57 | 56
Number analyzed (Woman years (rounded to nearest integer)) | 23 | 22
Pregnancies per 100 woman years | 0 [0 to 16.1] | 0 [0 to 17.1]

40. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding/Spotting
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: NOMAC-E2: 21-day period starting on Day 4 of the cycle; LNG-EE: 21-day period starting on Day 1 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n=number of participants with evaluable cycles.
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 18 | 16
  Cycle 2 (n=55 NOMAC-E2; n=51 LNG-EE) | 11 | 9
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 5 | 5
  Cycle 4 (n=54 NOMAC-E2; n=52 LNG-EE) | 8 | 2
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 6 | 4
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 6 | 3

41. Secondary Outcome: Number of Participants With an Occurrence of Absence of Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Absence of withdrawal bleeding was defined as no bleeding/spotting episode that began during or continued into the "expected bleeding period". Expected bleeding period: NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle; LNG-EE: 7-day period starting on Day 22 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 40
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 6 | 0
  Cycle 2 (n=55 NOMAC-E2; n=51 LNG-EE) | 8 | 1
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 5 | 0
  Cycle 4 (n=54 NOMAC-E2; n=52 LNG-EE) | 8 | 0
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 5 | 0
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 10 | 1

42. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding was defined as any bleeding episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: NOMAC-E2: 21-day period starting on Day 4 of the cycle; LNG-EE: 21-day period starting on Day 1 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 40
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 3 | 1
  Cycle 2 (n=55 NOMAC-E2; n=51 LNG-EE) | 1 | 0
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 1 | 0
  Cycle 4 (n=54 NOMAC-E2; n=52 LNG-EE) | 1 | 0
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 2 | 0
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 3 | 0

43. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Spotting (Spotting Only)
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough spotting was defined as any spotting episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: NOMAC-E2: 21-day period starting on Day 4 of the cycle; LNG-EE: 21-day period starting on Day 1 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 40
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 17 | 16
  Cycle 2 (n=55 NOMAC-E2; n=51 LNG-EE) | 10 | 9
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 4 | 5
  Cycle 4 (n=54 NOMAC-E2; n=52 LNG-EE) | 7 | 2
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 4 | 4
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 4 | 3

44. Secondary Outcome: Number of Participants With an Occurrence of Early Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Early withdrawal bleeding was defined as any withdrawal bleeding that started before the current "expected bleeding period". Expected bleeding period: NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle; LNG-EE: 7-day period starting on Day 22 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 40
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 5 | 4
  Cycle 2 (n=55 NOMAC-E2; n=51 LNG-EE) | 4 | 1
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 3 | 1
  Cycle 4 (n=54 NOMAC-E2; n=52 LNG-EE) | 2 | 0
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 1 | 0
  Cycle 6 (n=52 NOMAC-E2; n=50 LNG-EE) | 2 | 2

45. Secondary Outcome: Number of Participants With an Occurrence of Continued Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Continued withdrawal bleeding was defined as any withdrawal bleeding that continued into the "expected non-bleeding period" of the next cycle. Expected non-bleeding period: NOMAC-E2: 21-day period starting on Day 4 of the cycle; LNG-EE: 21-day period starting on Day 1 of the cycle.
Time Frame: Every 28-day cycle for 5 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
Measure: Number; unit: Participants
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 6 consecutive 28-day cycles.
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
- LNG-EE: Monophasic combined oral contraceptive (COC) tablets containing 0.150 mg levonorgestrel (LNG) and 0.030 mg
  ethinylestradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28 placebo tablets) for 6 consecutive 28-day cycles.
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Participants
  Cycle 1 (n=56 NOMAC-E2; n=53 LNG-EE) | 15 | 25
  Cycle 2 (n=54 NOMAC-E2; n=50 LNG-EE) | 11 | 28
  Cycle 3 (n=54 NOMAC-E2; n=52 LNG-EE) | 13 | 26
  Cycle 4 (n=53 NOMAC-E2; n=52 LNG-EE) | 11 | 27
  Cycle 5 (n=52 NOMAC-E2; n=51 LNG-EE) | 13 | 29

46. Secondary Outcome: Average Number of Breakthrough Bleeding/Spotting Days
Description: as for outcome 40
Time Frame: Every 28-day cycle for 6 cycles
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n=number of participants who had breakthrough bleeding/spotting for the respective cycle.
Measure: Mean (Standard Error); unit: Days
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Days
  Cycle 1 (n=18 NOMAC-E2; n=16 LNG-EE) | 3.5 (2.7) | 4.6 (3.6)
  Cycle 2 (n=11 NOMAC-E2; n=9 LNG-EE) | 4.3 (1.4) | 3.3 (2.2)
  Cycle 3 (n=5 NOMAC-E2; n=5 LNG-EE) | 4.6 (2.5) | 3.2 (2.2)
  Cycle 4 (n=8 NOMAC-E2; n=2 LNG-EE) | 3.8 (2.3) | 4.0 (0.0)
  Cycle 5 (n=6 NOMAC-E2; n=4 LNG-EE) | 3.3 (2.5) | 2.0 (2.0)
  Cycle 6 (n=6 NOMAC-E2; n=3 LNG-EE) | 4.7 (3.7) | 3.0 (2.0)

47. Secondary Outcome: Average Number of Withdrawal Bleeding/Spotting Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Withdrawal bleeding/spotting was defined as any episode that occurred during the "expected bleeding period". Expected bleeding period: NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle; LNG-EE: 7-day period starting on Day 22 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n=number of participants who had withdrawal bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 53
Days
  Cycle 1 (n=50 NOMAC-E2; n=53 LNG-EE) | 4.8 (2.3) | 5.8 (3.6)
  Cycle 2 (n=47 NOMAC-E2; n=50 LNG-EE) | 4.7 (3.6) | 4.9 (1.2)
  Cycle 3 (n=49 NOMAC-E2); n=52 LNG-EE) | 3.9 (2.0) | 4.9 (1.4)
  Cycle 4 (n=46 NOMAC-E2; n=52 LNG-EE) | 4.0 (2.5) | 5.0 (1.5)
  Cycle 5 (n=47 NOMAC-E2; n=51 LNG-EE) | 3.8 (1.7) | 4.9 (1.5)
  Cycle 6 (n=42 NOMAC-E2; n=49 LNG-EE) | 3.5 (1.2) | 4.2 (1.7)

ADVERSE EVENTS:
Arm/Group | NOMAC-E2 | LNG-EE
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/58
Other Adverse Events (participants affected / at risk) | 9/60 | 18/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=60) | LNG-EE (N=58)
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=60) | LNG-EE (N=58)
Influenza (Infections and infestations) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (14) | 5 (6)
Headache (Nervous system disorders) | 3 (5) | 7 (14)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the SPONSOR. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the SPONSOR, at least six weeks ahead of estimated publication or presentation, for consent, which shall not be withheld unreasonably.